CLINICAL TRIAL: NCT00543777
Title: Validation Study of Magnetic Resonance Elastography and 2-Point Dixon MR Imaging Techniques in Diffuse Liver Disease
Brief Title: Magnetic Resonance Elastography and 2-Point Dixon MR Imaging Techniques in Diffuse Liver Disease
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2007-0107; NCI-2011-00492 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2007-10-12; First posted 2007-10-15 (Estimated); Results first posted 2021-04-13 (Actual); Last update posted 2021-04-13 (Actual); Status verified 2021-03

CONDITIONS: Liver Cancer
Keywords: Liver Cancer; Magnetic Resonance Elastography; 2-Point Dixon Magnetic Resonance Imaging; Liver Disease; Fatty Liver; Liver Fibrosis; Liver Cirrhosis; MRE; 2PD MRI; phase correction algorithm
MeSH Terms: conditions — Liver Neoplasms; Liver Diseases; Fatty Liver; Liver Cirrhosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- MRE + 2PD MRI (Experimental): MRE - Pneumatic driver will be placed over the upper abdomen. Patient will feel a vibration (like a cell phone or beeper vibrating). This vibration will create very small waves in the body. The scanner will then receive the vibrations from the liver and use them to create images of the liver tissue. 2PD MRI - Imaging performed after the MRE procedure and lasting 20-60 seconds. This procedure is useful in identifying fat tissue.
  Interventions: Diagnostic Test: Magnetic Resonance Elastogram; Diagnostic Test: 2-Point Dixon Magnetic Resonance Imaging

INTERVENTIONS:
Diagnostic Test: Magnetic Resonance Elastogram — Pneumatic driver will be placed over the upper abdomen. Patient will feel a vibration (like a cell phone or beeper vibrating). This vibration will create very small waves in the body. The scanner will then receive the vibrations from the liver and use them to create images of the liver tissue.
  Other Names: MRE
Diagnostic Test: 2-Point Dixon Magnetic Resonance Imaging — Imaging performed after the MRE procedure and lasting 20-60 seconds. This procedure is useful in identifying fat tissue.
  Other Names: 2PD MRI

SUMMARY:
The goal of this clinical research study is to test the accuracy of magnetic resonance elastogram (MRE) and 2-point dixon magnetic resonance imaging (2PD MRI) using new computer software (called "phase correction algorithm") in patients who might have liver disease.

DETAILED DESCRIPTION:
Finding liver damage as early as possible is important. Traditionally, biopsies have been used for this purpose. Biopsies are accurate but can only check a small part of the liver. Tissue fat and liver stiffness are common in patients with liver disease.This study is testing new MRI techniques (called an MRE) that may be able to test for these symptoms on the entire liver, in a short time.

A typical MRI uses a large magnet instead of x-rays to take pictures of the inside of your body. The MRE will be done on a standard MRI scanner.

Study Visit:

The MRE procedure is useful for identifying tissue stiffness. For the MRE procedure, you will lie on your back on the examination table, and a pneumatic driver (a light-weight, clear plastic drum, about 10 inches wide and 1 inch thick) will be placed over the upper abdomen. You will feel a vibration (like a cell phone or beeper vibrating). This vibration will create very small waves in the body. The scanner will then receive the vibrations from the liver and use them to create images of the liver tissue. The MRE will take about 40 seconds. The driver will only be turned on during this time.

Once the MRE is completed, you will then have a 2PD MRI scan while you are still lying on the table. This procedure is useful in identifying fat tissue. This will take about 20-60 seconds. The total exam time will be no more than 20 minutes, including the preparation time.

Once the MRI is completed, you will have a liver biopsy as part of your standard care. You will sign a separate consent form for this procedure.

After the biopsy is performed, your participation in the study will be complete.

This is an investigational study. The scanners and software for 2PD MRI used for this study are FDA-approved and being used in clinical practice. The MRE technique used for this study has not been FDA-approved. At this time, the MRE technique is being used in research only. The use of study data for the purpose of this study is investigational. Up to 60 patients will take part in this study. All will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Group 1. Non-oncologic patients from VAMC in Houston:
2. Biopsy proven or clinically suspected advanced parenchymal liver disease
3. Core biopsies obtained within 1-month of MRI/MRE
4. No treatment affecting the status of liver between MRI/MRE and post-imaging biopsy
5. Signed consent
6. Group 2. Oncologic patients at MDACC:
7. Clinically or radiographically suspected liver damage, hepatic steatosis, hepatitis, hepatic fibrosis or cirrhosis
8. Surgical or core biopsy scheduled within 4 weeks of MRI/MRE
9. Signed consent

Exclusion Criteria:

1. Claustrophobia
2. Contraindications for MRI
3. Unable to hold a breath
4. Ascites or other clinical or radiographical signs of portal hypertension

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2007-09 (Actual); Primary Completion 2020-01-13 (Actual); Study Completion 2020-01-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Haesun Choi, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | MRE + 2PD MRI
Started | 44
Completed | 44
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | MRE + 2PD MRI
Number analyzed (Participants) | 44
Age, Continuous [Median (Full Range); unit: years] | 47 [38 to 53]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17
  Male | 27
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 44

OUTCOME MEASURES:

1. Primary Outcome: Overall Image Quality of Magnetic Resonance Elastography (MRE)
Time Frame: 2 Years
Population: MRE Data processing not conducted, therefore data could not be generated.
Arm/Group | MRE + 2PD MRI
Number analyzed (Participants) | 0

2. Secondary Outcome: Association Between Degrees of Stiffness Measured by MRE in kPa and Histopathological Grades of Fibrosis and Steatohepatitis
Description: Assessed using Pearson correlation
Time Frame: Baseline to end of trial, up to 2 years
Population: Association between degrees of stiffness measured by MRE in kPa and histopathological grades of fibrosis and steatohepatitis processing not conducted, therefore data could not generated.
Arm/Group | MRE + 2PD MRI
Number analyzed (Participants) | 0

3. Secondary Outcome: Hepatic Steatosis
Description: Development of a non-invasive means to quantify hepatic steatosis using 2-Point Dixon technique for patients with >30% steatosis compared to participants with <30% steatosis. The degree of steatosis was quantified by percent fat fraction (%FF).
Time Frame: Baseline to the end of the trial, up to 2 years
Population: Participants analyzed are those with liver tumors requiring hepatic resection.
Measure: Mean (Standard Deviation); unit: percentage of fat fraction
Arm/Group | MRE + 2PD MRI
Number analyzed (Participants) | 28
percentage of fat fraction
  >30% Steatosis | 22 (5.2)
  <30% Steatosis | 5.0 (2.1)

ADVERSE EVENTS:
Time Frame: Baseline to end of trial, up to 2 years
Arm/Group | MRE + 2PD MRI
All-Cause Mortality (participants affected / at risk) | 0/44
Serious Adverse Events (participants affected / at risk) | 0/44
Other Adverse Events (participants affected / at risk) | 0/44

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-02-12): https://cdn.clinicaltrials.gov/large-docs/77/NCT00543777/Prot_SAP_000.pdf